CLINICAL TRIAL: NCT04552925
Title: The Effectiveness of Exercises with Electromyographic Biofeedback in Conservative Treatment of Massive Rotator Cuff Tears: a Randomized Controlled Study
Brief Title: Exercises with Electromyographic Biofeedback in Conservative Treatment of Massive Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Pelin Tiryaki, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/1507
Record Dates: First submitted 2020-09-12; First posted 2020-09-17 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Rotator Cuff Tears
Keywords: massive rotator cuff tear; deltoid; electromyographic biofeedback; rehabilitation; nonoperative management
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Active Comparator): Exercise group will receive ROM exercises, stretching and anterior deltoid re-education exercises described by Levy et al. Subjects will treated at the clinic three times per week for 6 weeks (18 sessions).
  Interventions: Other: Rehabilitation
- EMG-BF Group (Experimental): EMG-BF group will receive the same exercises as with the other group, but deltoid re-education exercises were performed under the guidance of EMG-BF device. All subjects will treated at the clinic three times per week for 6 weeks (18 sessions).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Exercises and rehabilitation for massive rotator cuff tears

SUMMARY:
There are very few studies in the literature about conservative treatment of massive rotator cuff (RC) tears. Whether the treatment of massive RC tears is conservative or surgical is decided according to the age, activity level, expectation and additional pathologies of the patient. The aim of conservative treatment is to make the patient functionally independent and to reduce pain. In recent years, there are different opinions in the literature about the effectiveness of conservative treatment of massive RC tears. However, in recent biomechanical studies, it has been reported that the RC and the deltoid, which remain intact in massive RC tears, can function well together.

The hypothesis of this study is that the deltoid-focused physiotherapy program, where strengthening exercises are performed with EMG biofeedback, will give more positive results in terms of range of motion (ROM), functional status, muscle strength, pain and patients satisfaction. aim of our study is to investigate the efficacy of electromyographic biofeedback (EMG-BF) device which was added to deltoid focused conservative treatment program in massive RC tears.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, non-traumatic massive rotator cuff tears according to Deorio and Cofield classification
* Age older than 50 years and attend 1-year follow-up assessment

Exclusion Criteria:

* Patients with symptomatic lesions in the contralateral shoulder
* Cuff tear arthropathy
* Glenohumeral osteoarthritis
* Pseudoparalytic shoulder
* Grade 3-4 fatty degeneration according to Goutallier classification
* History of involved shoulder surgery
* Major systemic conditions that disallowing exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
American shoulder and elbow (ASES) score | 12 months
  The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) is a standard shoulder assessment form, which is comprised of objective and subjective sections and prepared by shoulder and elbow surgeons.
Deltoid Strength | 12 months
  Measurement of the strength of the deltoid muscle with a digital dynamometer.

SECONDARY OUTCOMES:
Range of Motion (ROM) | 12 months
  Active ROM will evaluate with a universal goniometer.
Numeric Pain Rating Scale (NPRS) | 12 months
  Participants' level of pain will assess by numeric pain rating scale (NPRS).
Global rating of change scale (GRCS) | 12 months
  The global rating of change scale (GRCS) which is five-point Likert scale will be use to evaluate the difference between the participants' health status from their perspective. It is ranging from -2 (very much worse), through 0 (unchanged) to +2 (much better).

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çelik, Professor, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiryaki P, Celik D, Bilsel K, Ersen A. Effectiveness of Exercises With Electromyographic Biofeedback in Conservative Treatment of Massive Rotator Cuff Tears: A Randomized Controlled Study. Am J Phys Med Rehabil. 2023 May 1;102(5):419-426. doi: 10.1097/PHM.0000000000002111. Epub 2022 Sep 23. PMID 36166658